CLINICAL TRIAL: NCT01134055
Title: MD7110852, A Phase 2b Dose-Ranging Study of Pazopanib Eye Drops Versus Ranibizumab Intravitreal Injections for the Treatment of Neovascular Age-Related Macular Degeneration
Brief Title: Dose Ranging Study of Pazopanib to Treat Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110852
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-12

CONDITIONS: Macular Degeneration
Keywords: ranibizumab; wet AMD; MD7110852; age related macular degeneration; age-related macular degeneration; macular degeneration; pazopanib
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- investigational arm 1 (Experimental): 5 mg/mL pazopanib eye drops TID with allowance for as-needed ranibizumab injection
  Interventions: Drug: pazopanib eye drops
- investigational arm 2 (Experimental): 5 mg/mL pazopanib eye drops QID with allowance for as-needed ranibizumab injection
  Interventions: Drug: pazopanib eye drops
- investigational arm 3 (Experimental): 10 mg/mL pazopanib eye drops BID with allowance for as-needed ranibizumab injection
  Interventions: Drug: pazopanib eye drops
- investigational arm 4 (Experimental): 10 mg/mL pazopanib eye drops TID with allowance for as-needed ranibizumab injection
  Interventions: Drug: pazopanib eye drops
- investigational arm 5 (Experimental): 10 mg/mL pazopanib eye drops QID with allowance for as-needed ranibizumab injection
  Interventions: Drug: pazopanib eye drops
- placebo control arm (Placebo Comparator): Placebo eye drops QID with allowance for as-needed ranibizumab injection
  Interventions: Drug: placebo
- active open-label control arm (Active Comparator): Ranibizumab intravitreal injection every 4 weeks
  Interventions: Biological: ranibizumab intravitreal injection

INTERVENTIONS:
Drug: pazopanib eye drops — A tyrosine kinase inhibitor of multiple receptors including vascular endothelial growth factor receptors and platelet-derived growth factor receptors.
  Arms: investigational arm 1; investigational arm 2; investigational arm 3; investigational arm 4; investigational arm 5
Drug: placebo — placebo eye drops
  Arms: placebo control arm
Biological: ranibizumab intravitreal injection — Humanized recombinant monoclonal antibody fragment targeted against human vascular endothelial growth factor A
  Arms: active open-label control arm

SUMMARY:
The purpose of this study is to determine the safety and efficacy of different dosage regimens of pazopanib eye drops for the treatment of neovascular age-related macular degeneration.

DETAILED DESCRIPTION:
MD7110852 is a Phase 2b dose-ranging study designed to demonstrate the 1 year efficacy and safety of pazopanib eye drops for the treatment of neovascular age related macular degeneration (AMD) in subjects whose disease is currently managed with anti-VEGF (vascular endothelial growth factor) injection therapy. Eye drop regimens are double-masked with placebo eye drops and will have access to open-label ranibizumab intravitreal (IVT) injection if needed. The ranibizumab IVT injection every 4 weeks control arm is open-label.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥50 years.
* Active subfoveal choroidal neovascularization (CNV) lesion secondary to AMD in study eye: Total lesion area ≤12 disc areas with CNV ≥50% total lesion area.
* Anti-Vascular endothelial growth factor (VEGF) intravitreal injection experienced and in need of re-treatment.
* Best-corrected visual acuity of at least 24 letters (equates to approximately 20/320 Snellen equivalents or better).

Exclusion Criteria:

* Prior ocular investigational drug/device for choroidal neovascularization, photodynamic therapy, radiation, subfoveal or juxtafoveal focal laser photocoagulation.
* Prior failure to anti-VEGF intravitreal injection therapy.
* Recent ocular investigational drug/device for non-CNV condition.
* Prior ocular surgeries (vitrectomy, scleral buckle, or glaucoma filtering/shunt surgery). Cataract surgery permitted if ≥3 months and has posterior chamber intraocular lens.
* Center-fovea involvement of any of the following: fibrosis, atrophy, serous retinal pigment epithelial detachment, or retinal pigment epithelial tear.
* CNV in either eye due to other causes.
* Clinical evidence of diabetic retinopathy or diabetic macular edema.
* Recent myocardial infarction or cerebrovascular accident.
* Uncontrolled hypertension in spite of antihypertensive medications.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2012-10-01 (Actual); Study Completion 2012-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (69):
- United States (34):
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Winter Haven, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Leawood, Kansas
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Beachwood, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Ashland, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Silverdale, Washington
  - GSK Investigational Site, Madison, Wisconsin
- Australia (3):
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
- Canada (6):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Toronto, Ontario
- Denmark (2):
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Glostrup Municipality
- Germany (7):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Kiel, Schleswig-Holstein
- Italy (4):
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Padua, Veneto
- Japan (7):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Tokyo
- Sweden (4):
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, randomized, parallel-group, double-masked eye drops, and active-controlled study from 01 June 2010 to 05 October 2012. The study was conducted at 77 sites in 9 countries from North America, Europe, Australia and Japan.
Pre-assignment Details: A total of 510 participants were randomized for the study. After a 1-2 week screening period, participants entered a 52-week treatment period. There were 449 screen failures in this study.
Groups:
- Placebo Control Arm QID: Only the study eye (one eye) per participant enrolled in the study received Placebo QID. Participants in this treatment arm were educated on the packaging and labeling of the eye drop, required refrigerated storage conditions, and proper dosing method. The study staff witnessed participants self-administering the first dose of the eye drop. Caregiver assistance was permitted. This witnessed dose occurred in the clinic on Day 1 of treatment. Participants continued to administer the eye drop daily for the duration of the 52-week treatment period. Ranibizumab IP injection was given whenever re-injection was necessary throughout the study.
- Pazopanib Eye Drops 5 mg/mL TID: Only the study eye (one eye) per participant enrolled in the study received pazopanib eye drops 5 milligram/milliliter (mg/mL) TID. Participants in this treatment arm were educated on the packaging and labeling of the eye drop, required refrigerated storage conditions, and proper dosing method. The study staff witnessed participants self-administering the first dose of the eye drop. Caregiver assistance was permitted. This witnessed dose occurred in the clinic on Day 1 of treatment. Participants continued to administer the eye drop daily for the duration of the 52-week Treatment Period. Ranibizumab IP injection was given whenever re-injection was necessary throughout the study.
- Pazopanib Eye Drops 5 mg/mL QID: Only the study eye (one eye) per participant enrolled in the study received pazopanib eye drops 5 mg/mL QID. Participants in this treatment arm were educated on the packaging and labeling of the eye drop, required refrigerated storage conditions, and proper dosing method. The study staff witnessed participants self-administering the first dose of the eye drop. Caregiver assistance was permitted. This witnessed dose occurred in the clinic on Day 1 of treatment. Participants continued to administer the eye drop daily for the duration of the 52-week Treatment Period. Ranibizumab IP injection was given whenever re-injection was necessary throughout the study.
- Pazopanib Eye Drops 10 mg/mL BID: Only the study eye (one eye) per participant enrolled in the study received pazopanib eye drops 10 mg/mL twice daily. Participants in this treatment arm were educated on the packaging and labeling of the eye drop, required refrigerated storage conditions, and proper dosing method. The study staff witnessed participants self-administering the first dose of the eye drop. Caregiver assistance was permitted. This witnessed dose occurred in the clinic on Day 1 of treatment. Participants continued to administer the eye drop daily for the duration of the 52-week Treatment Period. Ranibizumab IP injection was given whenever re-injection was necessary throughout the study.
- Pazopanib Eye Drops 10 mg/mL TID: Only the study eye (one eye) per participant enrolled in the study received pazopanib eye drops 10 mg/mL thrice daily. Participants in this treatment arm were educated on the packaging and labeling of the eye drop, required refrigerated storage conditions, and proper dosing method. The study staff witnessed participants self-administering the first dose of the eye drop. Caregiver assistance was permitted. This witnessed dose occurred in the clinic on Day 1 of treatment. Participants continued to administer the eye drop daily for the duration of the 52-week Treatment Period. Ranibizumab IP injection was given whenever re-injection was necessary throughout the study.
- Pazopanib Eye Drops 10 mg/mL QID: Only the study eye (one eye) per participant enrolled in the study received pazopanib eye drops 10 mg/mL four times daily. Participants in this treatment arm were educated on the packaging and labeling of the eye drop, required refrigerated storage conditions, and proper dosing method. The study staff witnessed participants self-administering the first dose of the eye drop. Caregiver assistance was permitted. This witnessed dose occurred in the clinic on Day 1 of treatment. Participants continued to administer the eye drop daily for the duration of the 52-week Treatment Period. Ranibizumab IP injection was given whenever re-injection was necessary throughout the study.
- Ranibizumab Injections Active Open-label Control Arm: Participants enrolled in this arm received no eye drops. They received a 0.20 mL to 0.23 mL fill of 10 mg/mL Ranibizumab injection once every four weeks throughout the entire 52 weeks of the study.
Period: Overall Study
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Started | 73 | 72 | 74 | 73 | 73 | 72 | 73
Completed | 65 | 66 | 71 | 67 | 67 | 65 | 62
Not Completed | 8 | 6 | 3 | 6 | 6 | 7 | 11
Not completed — Adverse Event | 5 | 2 | 2 | 2 | 5 | 7 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 1 | 2 | 0 | 0 | 8
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pazopanib Eye Drops 5 mg/mL TID: Only the study eye (one eye) per participant enrolled in the study received pazopanib eye drops 5 mg/mL TID. Participants in this treatment arm were educated on the packaging and labeling of the eye drop, required refrigerated storage conditions, and proper dosing method. The study staff witnessed participants self-administering the first dose of the eye drop. Caregiver assistance was permitted. This witnessed dose occurred in the clinic on Day 1 of treatment. Participants continued to administer the eye drop daily for the duration of the 52-week Treatment Period. Ranibizumab IP injection was given whenever re-injection was necessary throughout the study.
- Total: Total of all reporting groups
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm | Total
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73 | 510
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.6 (9.42) | 74.4 (7.60) | 75.1 (8.19) | 75.4 (8.42) | 75.6 (8.71) | 76.2 (8.00) | 74.9 (7.27) | 75.3 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 43 | 42 | 45 | 40 | 46 | 41 | 296
  Male | 34 | 29 | 32 | 28 | 33 | 26 | 32 | 214
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 4 | 5 | 6 | 5 | 4 | 6 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 68 | 67 | 69 | 67 | 68 | 68 | 67 | 474
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) as Measured by the Number of Letters Read on the Early Treatment of Diabetic Retinopathy Study (ETDRS) Grading Charts at a Starting Distance of 4 Meters at Week 52
Description: BCVA was measured in the study eye using the ETDRS grading charts starting at a test distance of 4 meters. The ETDRS grading chart was of at least 24 to 78 letters. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. There were seven cut off points in change from baseline visual acuity on ETDRS grading chart which are, 15 to 29, 10 to 14, 5 to 9, -4 to 4, -5 to -9, -10 to -14 and -15 to -29 letters. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. If either the baseline or post-randomization value was missing, the change from baseline was set to missing as well. Day 1 values are considered as Baseline in this study.
Time Frame: Day 1 and 52 weeks
Population: Intent to Treat Population - It consisted of all randomized participants, according to the treatment groups assigned by randomization (i.e., planned rather than the actual treatment regimen), who received at least one dose of study medication. Only participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Letters
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Letters | 0.22 (1.006) | 1.15 (1.004) | 1.81 (0.975) | 0.76 (0.995) | 0.28 (0.992) | 0.62 (1.007) | 1.42 (1.020)

2. Secondary Outcome: Percentage of Ranibizumab Re-injections Received Over 28 and 52 Weeks
Description: The investigator interpreted each Week 4 to Week 52 Optical coherence tomography (OCT) scan, BCVA score, and available Fluorescein angiography (FA)/Fundus photography (FP) and re-injected if one or more criteria were met. The criteria were: Evidence of Intraretinal (IR) (with or without cysts) fluid or Subretinal (SR) fluid, a serous retinal pigment epithelial detachment, a notable decline in Visual Acuity, new SR or IR macular hemorrhage that the investigator judges is associated with Choroidal neovascularization, increased lesion size on FA relative to the last angiogram as judged by the investigator or leakage on FA that the investigator judges would benefit from re-injection. Injection rate over 52 weeks was computed by taking the number of injections received divided by the number of visits for the participant. Likewise for 28 weeks it was estimated as the number of post baseline injections received divided by the number of post baseline visits at or before the week 28 visit.
Time Frame: Up to 52 weeks
Population: Intent to Treat Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of re-injections
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72
Percentage of re-injections
  Injection Rate at 28 Weeks | 65.04 (3.418) | 55.03 (3.441) | 67.92 (3.395) | 66.11 (3.418) | 61.61 (3.418) | 59.42 (3.441)
  Overall Injection Rate at 52 weeks | 64.24 (3.263) | 55.09 (3.286) | 65.87 (3.241) | 62.50 (3.263) | 64.42 (3.263) | 58.19 (3.286)
Statistical Analysis 1: Comparison: Placebo Control Arm QID vs Pazopanib Eye Drops 5 mg/mL TID; Statistics for Injection Rate at 28 Weeks is presented; Test type: Superiority or Other; p = 0.1974, ANOVA — Adjusted p-Value has been presented
Statistical Analysis 2: Comparison: Placebo Control Arm QID vs Pazopanib Eye Drops 5 mg/mL QID; Statistics for Injection Rate at 28 Weeks is presented; Test type: Superiority or Other; p = 0.8263, ANOVA — Adjusted p-Value has been presented
Statistical Analysis 3: Comparison: Placebo Control Arm QID vs Pazopanib Eye Drops 10 mg/mL BID; Statistics for Injection Rate at 28 Weeks is presented; Test type: Superiority or Other; p = 0.8263, ANOVA — Adjusted p-Value has been presented
Statistical Analysis 4: Comparison: Placebo Control Arm QID vs Pazopanib Eye Drops 10 mg/mL TID; Statistics for Injection Rate at 28 Weeks is presented; Test type: Superiority or Other; p = 0.8263, ANOVA — Adjusted p-Value has been presented
Statistical Analysis 5: Comparison: Placebo Control Arm QID vs Pazopanib Eye Drops 10 mg/mL QID; Statistics for Injection Rate at 28 Weeks is presented; Test type: Superiority or Other; p = 0.7418, ANOVA — Adjusted p-Value has been presented
Statistical Analysis 6: Comparison: Placebo Control Arm QID vs Pazopanib Eye Drops 5 mg/mL TID; Statistics for Overall Injection Rate at 52 weeks is presented; Test type: Superiority or Other; p = 0.2429, ANOVA — Adjusted p-Value has been presented
Statistical Analysis 7: Comparison: Placebo Control Arm QID vs Pazopanib Eye Drops 5 mg/mL QID; Statistics for Overall Injection Rate at 52 weeks is presented; Test type: Superiority or Other; p = 0.9700, ANOVA — Adjusted p-Value has been presented
Statistical Analysis 8: Comparison: Placebo Control Arm QID vs Pazopanib Eye Drops 10 mg/mL BID; Statistics for Overall Injection Rate at 52 weeks is presented; Test type: Superiority or Other; p = 0.9700, ANOVA — Adjusted p-Value has been presented
Statistical Analysis 9: Comparison: Placebo Control Arm QID vs Pazopanib Eye Drops 10 mg/mL TID; Statistics for Overall Injection Rate at 52 weeks is presented; Test type: Superiority or Other; p = 0.9700, ANOVA — Adjusted p-Value has been presented
Statistical Analysis 10: Comparison: Placebo Control Arm QID vs Pazopanib Eye Drops 10 mg/mL QID; Statistics for Overall Injection Rate at 52 weeks is presented; Test type: Superiority or Other; p = 0.7673, ANOVA — Adjusted p-Value has been presented

3. Secondary Outcome: Number of Participants With BCVA Over Time
Description: BCVA was measured in the study eye using the ETDRS grading charts starting at a test distance of 4 meters. The ETDRS grading chart was of at least 24 to 78 letters. There were seven cut off points in change from baseline visual acuity on ETDRS grading chart which are, 15 to 29, 10 to 14, 5 to 9, -4 to 4, -5 to -9, -10 to -14 and -15 to -29 letters.
Time Frame: Up to Week 52
Population: Intent to Treat Population. Only participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Pazopanib Eye Drops 10 mg/mL BID: Only the study eye (one eye) per participant enrolled in the study received 10 mg/mL twice daily. Participants in this treatment arm were educated on the packaging and labeling of the eye drop, required refrigerated storage conditions, and proper dosing method. The study staff witnessed participants self-administering the first dose of the eye drop. Caregiver assistance was permitted. This witnessed dose occurred in the clinic on Day 1 of treatment. Participants continued to administer the eye drop daily for the duration of the 52-week Treatment Period. Ranibizumab IP injection was given whenever re-injection was necessary throughout the study.
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Participants
  Week 4, Study Eye: number analyzed (Participants) | 71 | 71 | 74 | 72 | 73 | 71 | 73
  Week 4, Study Eye: within 5 letters | 49 | 49 | 57 | 57 | 58 | 57 | 62
  Week 4, Study Eye: within 10 letters | 11 | 15 | 12 | 13 | 12 | 11 | 8
  Week 4, Study Eye: within 15 letters | 6 | 5 | 5 | 1 | 3 | 2 | 3
  Week 4, Study Eye: more than 15 letters | 5 | 2 | 0 | 1 | 0 | 1 | 0
  Week 4, Fellow Eye: number analyzed (Participants) | 72 | 71 | 73 | 72 | 73 | 71 | 73
  Week 4, Fellow Eye: within 5 letters | 53 | 57 | 65 | 59 | 61 | 60 | 60
  Week 4, Fellow Eye: within 10 letters | 16 | 12 | 6 | 12 | 11 | 7 | 11
  Week 4, Fellow Eye: within 15 letters | 2 | 2 | 2 | 1 | 1 | 3 | 2
  Week 4, Fellow Eye: more than 15 letters | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Week 8, Study Eye: number analyzed (Participants) | 71 | 70 | 74 | 73 | 71 | 71 | 72
  Week 8, Study Eye: within 5 letters | 34 | 36 | 51 | 51 | 44 | 47 | 54
  Week 8, Study Eye: within 10 letters | 21 | 23 | 18 | 18 | 20 | 16 | 14
  Week 8, Study Eye: within 15 letters | 11 | 7 | 5 | 1 | 6 | 7 | 4
  Week 8, Study Eye: more than 15 letters | 5 | 4 | 0 | 3 | 1 | 1 | 0
  Week 8, Fellow Eye: number analyzed (Participants) | 72 | 70 | 73 | 73 | 71 | 71 | 72
  Week 8, Fellow Eye: within 5 letters | 42 | 48 | 60 | 52 | 52 | 55 | 51
  Week 8, Fellow Eye: within 10 letters | 19 | 17 | 10 | 20 | 18 | 11 | 15
  Week 8, Fellow Eye: within 15 letters | 9 | 5 | 2 | 1 | 1 | 3 | 5
  Week 8, Fellow Eye: more than 15 letters | 2 | 0 | 1 | 0 | 0 | 2 | 1
  Week 12, Study Eye: number analyzed (Participants) | 71 | 68 | 74 | 72 | 72 | 69 | 70
  Week 12, Study Eye: within 5 letters | 26 | 25 | 48 | 41 | 35 | 34 | 46
  Week 12, Study Eye: within 10 letters | 27 | 30 | 17 | 23 | 25 | 24 | 22
  Week 12, Study Eye: within 15 letters | 13 | 8 | 8 | 4 | 10 | 9 | 2
  Week 12, Study Eye: more than 15 letters | 5 | 5 | 1 | 4 | 2 | 2 | 0
  Week 12, Fellow Eye: number analyzed (Participants) | 72 | 68 | 73 | 71 | 72 | 69 | 70
  Week 12, Fellow Eye: within 5 letters | 36 | 41 | 52 | 46 | 47 | 49 | 45
  Week 12, Fellow Eye: within 10 letters | 23 | 18 | 18 | 20 | 23 | 16 | 18
  Week 12, Fellow Eye: within 15 letters | 9 | 8 | 2 | 4 | 2 | 1 | 6
  Week 12, Fellow Eye: more than 15 letters | 4 | 1 | 1 | 1 | 0 | 3 | 1
  Week 16, Study Eye: number analyzed (Participants) | 71 | 68 | 73 | 70 | 71 | 69 | 68
  Week 16, Study Eye: within 5 letters | 24 | 20 | 41 | 36 | 26 | 26 | 35
  Week 16, Study Eye: within 10 letters | 28 | 37 | 22 | 25 | 29 | 29 | 30
  Week 16, Study Eye: within 15 letters | 10 | 4 | 9 | 4 | 13 | 11 | 3
  Week 16, Study Eye: more than 15 letters | 9 | 7 | 1 | 5 | 3 | 3 | 0
  Week 16, Fellow Eye: number analyzed (Participants) | 72 | 68 | 72 | 70 | 71 | 69 | 68
  Week 16, Fellow Eye: within 5 letters | 35 | 32 | 47 | 40 | 42 | 43 | 39
  Week 16, Fellow Eye: within 10 letters | 24 | 24 | 21 | 25 | 25 | 20 | 19
  Week 16, Fellow Eye: within 15 letters | 9 | 8 | 3 | 4 | 4 | 3 | 7
  Week 16, Fellow Eye: more than 15 letters | 4 | 4 | 1 | 1 | 0 | 3 | 3
  Week 20, Study Eye: number analyzed (Participants) | 69 | 68 | 71 | 70 | 71 | 69 | 67
  Week 20, Study Eye: within 5 letters | 21 | 19 | 32 | 32 | 26 | 21 | 30
  Week 20, Study Eye: within 10 letters | 32 | 36 | 25 | 26 | 30 | 32 | 31
  Week 20, Study Eye: within 15 letters | 10 | 5 | 12 | 8 | 12 | 11 | 5
  Week 20, Study Eye: more than 15 letters | 6 | 8 | 2 | 4 | 3 | 5 | 1
  Week 20, Fellow Eye: number analyzed (Participants) | 70 | 68 | 70 | 69 | 71 | 69 | 67
  Week 20, Fellow Eye: within 5 letters | 28 | 28 | 41 | 34 | 32 | 40 | 35
  Week 20, Fellow Eye: within 10 letters | 28 | 27 | 25 | 28 | 33 | 23 | 20
  Week 20, Fellow Eye: within 15 letters | 10 | 9 | 3 | 4 | 6 | 3 | 8
  Week 20, Fellow Eye: more than 15 letters | 4 | 4 | 1 | 3 | 0 | 3 | 4
  Week 24, Study Eye: number analyzed (Participants) | 69 | 68 | 72 | 69 | 71 | 69 | 66
  Week 24, Study Eye: within 5 letters | 19 | 16 | 28 | 26 | 23 | 20 | 25
  Week 24, Study Eye: within 10 letters | 29 | 36 | 30 | 31 | 34 | 32 | 34
  Week 24, Study Eye: within 15 letters | 14 | 8 | 12 | 9 | 11 | 11 | 6
  Week 24, Study Eye: more than 15 letters | 7 | 8 | 2 | 3 | 3 | 6 | 1
  Week 24, Fellow Eye: number analyzed (Participants) | 70 | 68 | 71 | 69 | 71 | 69 | 66
  Week 24, Fellow Eye: within 5 letters | 27 | 24 | 36 | 32 | 32 | 36 | 33
  Week 24, Fellow Eye: within 10 letters | 30 | 29 | 29 | 25 | 30 | 25 | 22
  Week 24, Fellow Eye: within 15 letters | 8 | 11 | 5 | 9 | 9 | 3 | 7
  Week 24, Fellow Eye: more than 15 letters | 5 | 4 | 1 | 3 | 0 | 5 | 4
  Week 28, Study Eye: number analyzed (Participants) | 68 | 68 | 71 | 69 | 70 | 68 | 66
  Week 28, Study Eye: within 5 letters | 19 | 13 | 26 | 24 | 22 | 17 | 18
  Week 28, Study Eye: within 10 letters | 30 | 37 | 29 | 33 | 32 | 33 | 35
  Week 28, Study Eye: within 15 letters | 14 | 9 | 14 | 9 | 11 | 10 | 10
  Week 28, Study Eye: more than 15 letters | 5 | 9 | 2 | 3 | 5 | 8 | 3
  Week 28, Fellow Eye: number analyzed (Participants) | 69 | 68 | 70 | 68 | 70 | 68 | 66
  Week 28, Fellow Eye: within 5 letters | 26 | 24 | 34 | 27 | 29 | 34 | 31
  Week 28, Fellow Eye: within 10 letters | 29 | 30 | 27 | 27 | 33 | 27 | 22
  Week 28, Fellow Eye: within 15 letters | 7 | 10 | 7 | 9 | 7 | 2 | 6
  Week 28, Fellow Eye: more than 15 letters | 7 | 4 | 2 | 5 | 1 | 5 | 7
  Week 32, Study Eye: number analyzed (Participants) | 67 | 68 | 70 | 69 | 68 | 66 | 63
  Week 32, Study Eye: within 5 letters | 17 | 11 | 23 | 23 | 20 | 14 | 12
  Week 32, Study Eye: within 10 letters | 32 | 37 | 33 | 32 | 32 | 35 | 38
  Week 32, Study Eye: within 15 letters | 14 | 11 | 11 | 10 | 12 | 9 | 10
  Week 32, Study Eye: more than 15 letters | 4 | 9 | 3 | 4 | 4 | 8 | 3
  Week 32, Fellow Eye: number analyzed (Participants) | 68 | 68 | 69 | 69 | 68 | 66 | 63
  Week 32, Fellow Eye: within 5 letters | 23 | 23 | 30 | 24 | 27 | 30 | 24
  Week 32, Fellow Eye: within 10 letters | 31 | 31 | 31 | 30 | 34 | 26 | 25
  Week 32, Fellow Eye: within 15 letters | 8 | 10 | 5 | 8 | 4 | 5 | 6
  Week 32, Fellow Eye: more than 15 letters | 6 | 4 | 3 | 7 | 3 | 5 | 8
  Week 36, Study Eye: number analyzed (Participants) | 65 | 66 | 71 | 68 | 69 | 67 | 63
  Week 36, Study Eye: within 5 letters | 16 | 10 | 22 | 20 | 19 | 13 | 12
  Week 36, Study Eye: within 10 letters | 31 | 36 | 34 | 34 | 32 | 35 | 41
  Week 36, Study Eye: within 15 letters | 14 | 11 | 13 | 7 | 15 | 9 | 8
  Week 36, Study Eye: more than 15 letters | 4 | 9 | 2 | 7 | 3 | 10 | 2
  Week 36, Fellow Eye: number analyzed (Participants) | 67 | 66 | 70 | 68 | 69 | 67 | 63
  Week 36, Fellow Eye: within 5 letters | 22 | 19 | 29 | 21 | 25 | 26 | 21
  Week 36, Fellow Eye: within 10 letters | 31 | 31 | 32 | 34 | 38 | 32 | 27
  Week 36, Fellow Eye: within 15 letters | 6 | 12 | 6 | 8 | 3 | 4 | 7
  Week 36, Fellow Eye: more than 15 letters | 8 | 4 | 3 | 5 | 3 | 5 | 8
  Week 40, Study Eye: number analyzed (Participants) | 67 | 68 | 70 | 68 | 68 | 67 | 62
  Week 40, Study Eye: within 5 letters | 14 | 11 | 19 | 20 | 18 | 13 | 12
  Week 40, Study Eye: within 10 letters | 33 | 32 | 35 | 34 | 34 | 34 | 38
  Week 40, Study Eye: within 15 letters | 12 | 16 | 14 | 7 | 11 | 9 | 10
  Week 40, Study Eye: more than 15 letters | 8 | 9 | 2 | 7 | 5 | 11 | 2
  Week 40, Fellow Eye: number analyzed (Participants) | 68 | 68 | 69 | 68 | 67 | 67 | 63
  Week 40, Fellow Eye: within 5 letters | 20 | 16 | 23 | 21 | 23 | 25 | 21
  Week 40, Fellow Eye: within 10 letters | 31 | 36 | 37 | 35 | 35 | 33 | 28
  Week 40, Fellow Eye: within 15 letters | 9 | 13 | 6 | 7 | 5 | 3 | 5
  Week 40, Fellow Eye: more than 15 letters | 8 | 3 | 3 | 5 | 4 | 6 | 9
  Week 44, Study Eye: number analyzed (Participants) | 66 | 68 | 70 | 67 | 67 | 65 | 62
  Week 44, Study Eye: within 5 letters | 11 | 10 | 18 | 17 | 17 | 13 | 11
  Week 44, Study Eye: within 10 letters | 36 | 33 | 35 | 32 | 33 | 32 | 38
  Week 44, Study Eye: within 15 letters | 10 | 16 | 14 | 12 | 12 | 9 | 12
  Week 44, Study Eye: more than 15 letters | 9 | 9 | 3 | 6 | 5 | 11 | 1
  Week 44, Fellow Eye: number analyzed (Participants) | 67 | 68 | 69 | 67 | 67 | 65 | 63
  Week 44, Fellow Eye: within 5 letters | 15 | 16 | 22 | 20 | 21 | 25 | 19
  Week 44, Fellow Eye: within 10 letters | 35 | 36 | 36 | 32 | 36 | 30 | 29
  Week 44, Fellow Eye: within 15 letters | 8 | 12 | 7 | 9 | 6 | 4 | 7
  Week 44, Fellow Eye: more than 15 letters | 9 | 4 | 4 | 6 | 4 | 6 | 8
  Week 48, Study Eye: number analyzed (Participants) | 64 | 67 | 71 | 67 | 68 | 66 | 62
  Week 48, Study Eye: within 5 letters | 10 | 9 | 14 | 16 | 15 | 13 | 11
  Week 48, Study Eye: within 10 letters | 36 | 32 | 37 | 31 | 36 | 32 | 36
  Week 48, Study Eye: within 15 letters | 9 | 18 | 16 | 13 | 12 | 11 | 13
  Week 48, Study Eye: more than 15 letters | 9 | 8 | 4 | 7 | 5 | 10 | 2
  Week 48, Fellow Eye: number analyzed (Participants) | 65 | 67 | 70 | 66 | 68 | 66 | 62
  Week 48, Fellow Eye: within 5 letters | 14 | 14 | 20 | 18 | 21 | 24 | 17
  Week 48, Fellow Eye: within 10 letters | 35 | 36 | 40 | 33 | 38 | 31 | 26
  Week 48, Fellow Eye: within 15 letters | 8 | 12 | 5 | 8 | 7 | 5 | 10
  Week 48, Fellow Eye: more than 15 letters | 8 | 5 | 5 | 7 | 2 | 6 | 9
  Week 52, Study Eye: number analyzed (Participants) | 64 | 66 | 71 | 67 | 67 | 64 | 62
  Week 52, Study Eye: within 5 letters | 11 | 8 | 12 | 15 | 13 | 13 | 10
  Week 52, Study Eye: within 10 letters | 32 | 31 | 38 | 31 | 37 | 31 | 35
  Week 52, Study Eye: within 15 letters | 11 | 19 | 15 | 14 | 10 | 8 | 15
  Week 52, Study Eye: more than 15 letters | 10 | 8 | 6 | 7 | 7 | 12 | 2
  Week 52, Fellow Eye: number analyzed (Participants) | 64 | 66 | 70 | 67 | 67 | 64 | 61
  Week 52, Fellow Eye: within 5 letters | 13 | 14 | 20 | 19 | 18 | 21 | 16
  Week 52, Fellow Eye: within 10 letters | 35 | 35 | 39 | 31 | 38 | 33 | 28
  Week 52, Fellow Eye: within 15 letters | 8 | 11 | 5 | 9 | 9 | 5 | 10
  Week 52, Fellow Eye: more than 15 letters | 8 | 6 | 6 | 8 | 2 | 5 | 7

4. Secondary Outcome: Number of Participants Analyzed for Visual Acuity (VA) Response Over Time
Description: VA was measured in the study eye using the ETDRS grading charts starting at a test distance of 4 meters.The ETDRS grading chart was of at least 24 to 78 letters. There were seven cut off points in change from baseline visual acuity on ETDRS grading chart which are, 15 to 29, 10 to 14, 5 to 9, -4 to 4, -5 to -9, -10 to -14 and -15 to -29 letters. This outcome measure contains the number of participants who were analyzed for VA response.
Time Frame: Week 52
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Participants | 25 | 19 | 20 | 18 | 21 | 23 | 15

5. Secondary Outcome: Change From Baseline in Center Point Thickness (CPT) Over Time
Description: CPT was the inner limiting membrane to the beginning of the retinal pigment epithelium (RPE) inclusive of SR fluid. The outer boundary included the outer segment of the photoreceptors and not included the RPE. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. If either the baseline or post-randomization value was missing, the change from baseline was set to missing as well. Day 1 values are considered as Baseline in this study. In amendment 3, inclusion criterion number 5 was revised to remove the required quantitative OCT component. OCT examination was used to supplement FA findings and provided qualitative (presence of SR and/or IR fluid) and quantitative (a CPT that is at least 250 microns) evidence of an active subfoveal lesion. Hence data for pre and post amendment have been provided separately.
Time Frame: Baseline and Week 52
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Microns
  Subgroup-Genotype, Week 28, CC: number analyzed (Participants) | 22 | 19 | 21 | 25 | 18 | 22 | 21
  Subgroup-Genotype, Week 28, CC | 10.0 (55.29) | 12.3 (48.05) | 3.4 (56.23) | -27.6 (136.79) | 16.6 (75.36) | 9.7 (76.41) | -10.4 (79.28)
  Subgroup-Genotype, Week 28, CT: number analyzed (Participants) | 32 | 37 | 30 | 24 | 31 | 34 | 32
  Subgroup-Genotype, Week 28, CT | 9.6 (77.04) | 11.1 (62.94) | 9.4 (84.10) | -8.9 (54.05) | -8.4 (87.97) | 4.2 (72.25) | -18.1 (101.47)
  Subgroup-Genotype, Week 52, CC: number analyzed (Participants) | 21 | 19 | 21 | 23 | 16 | 21 | 21
  Subgroup-Genotype, Week 52, CC | 12.7 (76.07) | 6.9 (63.99) | 3.6 (95.68) | -37.3 (118.33) | 31.4 (56.63) | 7.4 (93.46) | -40.8 (72.12)
  Subgroup-Genotype, Week 52, CT: number analyzed (Participants) | 29 | 35 | 30 | 22 | 30 | 32 | 31
  Subgroup-Genotype, Week 52, CT | -2.9 (48.00) | 5.5 (73.67) | -10.5 (65.41) | -9.7 (61.55) | -12.3 (101.63) | -7.2 (89.75) | -14.2 (108.24)
  Subgroup-Pre-amendment 3, Week 28: number analyzed (Participants) | 8 | 12 | 12 | 10 | 11 | 12 | 12
  Subgroup-Pre-amendment 3, Week 28 | 20.9 (104.87) | 30.8 (75.58) | -15.9 (64.65) | -44.4 (114.54) | 27.8 (113.06) | -28.5 (101.42) | -16.6 (89.64)
  Subgroup-Post-amendment 3, Week 28: number analyzed (Participants) | 61 | 56 | 59 | 59 | 59 | 56 | 52
  Subgroup-Post-amendment 3, Week 28 | 9.9 (72.13) | 11.0 (53.06) | 8.5 (65.28) | -8.6 (92.03) | -7.7 (66.09) | 14.1 (65.43) | -15.0 (87.50)
  Subgroup-Pre-amendment 3, Week 52: number analyzed (Participants) | 7 | 12 | 12 | 9 | 10 | 12 | 11
  Subgroup-Pre-amendment 3, Week 52 | -24.1 (66.83) | 13.8 (120.91) | -57.8 (85.39) | -50.3 (63.87) | -8.2 (56.80) | -9.0 (142.59) | -29.0 (91.44)
  Subgroup-Post-amendment 3, Week 52: number analyzed (Participants) | 57 | 54 | 59 | 56 | 57 | 52 | 52
  Subgroup-Post-amendment 3, Week 52 | 0.1 (64.33) | 9.6 (61.19) | 2.2 (74.83) | -13.7 (97.67) | 3.2 (86.08) | -3.0 (67.15) | -23.5 (90.13)

6. Secondary Outcome: Number of Participants That Met Criteria for Re-injection
Description: The investigator interpreted each Week 4 to Week 52 Optical coherence tomography (OCT) scan, BCVA score, and available Fluorescein angiography (FA)/Fundus photography (FP) and re-injected if one or more criteria were met. The criteria were: Evidence of Intraretinal (IR) (with or without cysts) fluid or Subretinal (SR) fluid, a serous retinal pigment epithelial detachment, a notable decline in Visual Acuity, new SR or IR macular hemorrhage that the investigator judges is associated with Choroidal neovascularization, increased lesion size on FA relative to the last angiogram as judged by the investigator or leakage on FA that the investigator judges would benefit from re-injection.
Time Frame: Up to Week 52
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72
Participants
  Week 4: number analyzed (Participants) | 64 | 59 | 66 | 67 | 61 | 62
  Week 4 | 49 | 33 | 54 | 48 | 45 | 44
  Week 12: number analyzed (Participants) | 60 | 60 | 68 | 66 | 59 | 57
  Week 12 | 45 | 40 | 49 | 47 | 46 | 42
  Week 16: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0
  Week 16 | 1 | 0 | 0 | 0 | 0 | 0
  Week 20 | 0 | 0 | 0 | 1 | 0 | 0
  Week 28: number analyzed (Participants) | 54 | 58 | 62 | 60 | 56 | 50
  Week 28 | 38 | 41 | 45 | 47 | 39 | 36
  Week 32: number analyzed (Participants) | 73 | 72 | 74 | 1 | 73 | 1
  Week 32 | 0 | 0 | 0 | 1 | 0 | 1
  Week 44: number analyzed (Participants) | 73 | 1 | 74 | 73 | 73 | 72
  Week 44 | 0 | 1 | 0 | 0 | 0 | 0
  Week 52: number analyzed (Participants) | 50 | 52 | 61 | 55 | 52 | 54
  Week 52 | 36 | 28 | 43 | 37 | 45 | 36

7. Secondary Outcome: Change From Baseline in the Area of Choroidal Neovascularisation (CNV)
Description: Choroidal neovascularisation is progressive worsening of vision that can cause hemorrhage and exudation, and finally disciform scarring and retinal atrophy. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. If either the baseline or post-randomization value was missing, the change from baseline was set to missing as well. Day 1 values are considered as Baseline in this study.
Time Frame: Day 1, Week 28 and Week 52
Population: Intent to Treat Population
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)^2
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Millimeter (mm)^2
  Week 28 | 0.10 (0.113) | 0.16 (0.114) | 0.09 (0.111) | 0.06 (0.114) | -0.05 (0.112) | 0.13 (0.114) | -0.08 (0.118)
  Week 52 | 0.10 (0.134) | 0.13 (0.133) | 0.08 (0.129) | -0.16 (0.134) | -0.10 (0.132) | 0.13 (0.134) | -0.08 (0.137)

8. Secondary Outcome: Change From Baseline in the Area of the CNV Lesion Complex (i.e. CNV, Blood, PED, and Fibrosis)
Description: CNV is progressive worsening of vision that can cause hemorrhage and exudation, and finally disciform scarring and retinal atrophy. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. If either the baseline or post-randomization value was missing, the change from baseline was set to missing as well. Day 1 values are considered as Baseline in this study.
Time Frame: Day 1, Week 28 and Week 52
Population: Intent to Treat Population
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
mm^2
  Week 28 | 0.18 (0.131) | 0.32 (0.132) | 0.23 (0.129) | 0.12 (0.132) | 0.00 (0.130) | 0.13 (0.132) | -0.13 (0.137)
  Week 52 | 0.40 (0.152) | 0.51 (0.151) | 0.09 (0.146) | 0.01 (0.151) | -0.05 (0.150) | 0.20 (0.152) | -0.11 (0.155)

9. Secondary Outcome: Change From Baseline in the Area of Fluorescein Leakage
Description: Fluorescein angiograms was performed at the Screening, Week 12, Week 28, and Week 52 Visits. All images, including any that were performed at the investigator's medical discretion, were transferred to the FPRC. Fluorescein was injected intravenously according to usual clinic procedures. Dose response was also examined under different aspects of re-injection, such as time to first injection, the percentage of participants that required an injection by Week 28, as well as the estimation of the probability of reinjection. FA assessments of area of fluorescein leakage, CNV area and area of CNV lesion complex were also examined for dose differentiation.
Time Frame: Day 1, Week 28 and Week 52
Population: Intent to Treat Population
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
mm^2
  Week 28 | -0.33 (0.150) | -0.27 (0.151) | -0.32 (0.148) | -0.40 (0.151) | -0.61 (0.149) | -0.33 (0.151) | -0.60 (0.156)
  Week 52 | -0.40 (0.177) | -0.45 (0.176) | -0.19 (0.171) | -0.77 (0.177) | -0.57 (0.175) | -0.37 (0.178) | -0.66 (0.181)

10. Secondary Outcome: Change in Area of Serous Sensory Retinal Detachment (SSRD)
Description: This is an Optical coherence tomography (OCT) parameter used to manually measure thickness along any scan. OCT was performed at week 28 and week 52.
Time Frame: Day 1, Week 28 and Week 52
Population: Intent to Treat Population
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
mm^2
  Week 28 | -0.30 (0.259) | -0.28 (0.264) | -0.14 (0.255) | -0.55 (0.261) | -0.64 (0.261) | -0.46 (0.264) | -0.95 (0.273)
  Week 52 | -0.52 (0.317) | -0.76 (0.315) | -0.79 (0.300) | -1.24 (0.312) | -1.17 (0.321) | -0.83 (0.321) | -1.02 (0.322)

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Up to 52 Weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Participants
  Adverse Events (AEs) | 11 | 10 | 12 | 11 | 10 | 11 | 6
  Serious Adverse Events (SAEs) | 52 | 34 | 47 | 44 | 46 | 41 | 42

12. Secondary Outcome: Summary of Potentially Clinically Important Findings for Ophthalmic Examinations
Description: Opthalmicexaminations were done on Ocular alignment and motility, pupillary function, and visual fields by confrontation. Slit-lamp biomicroscopic examination of the anterior segment structure was performed. Fundus slit-lamp biomicroscopic examination, including use of accessory diagnostic lenses, to view the vitreous, retina (including posterior pole and periphery), macula, vasculature, and optic nerve was also performed. These examinations were performed on the study eye (SE) and the Fellow eye (FE). Participants with abnormal findings are listed here.
Time Frame: Up to Week 52
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Participants
  Afferent papillary defect present, SE | 4 | 2 | 4 | 2 | 1 | 2 | 3
  Afferent papillary defect present, FE | 4 | 1 | 5 | 2 | 3 | 2 | 3
  Eye motility abnormal, SE | 1 | 0 | 0 | 1 | 0 | 0 | 1
  Eye motility abnormal, FE | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Confrontation visual field abnormal, SE | 2 | 1 | 0 | 0 | 0 | 1 | 0
  Confrontation visual field abnormal, FE | 2 | 0 | 2 | 1 | 2 | 0 | 2
  Ptosis present, SE | 2 | 1 | 1 | 0 | 8 | 2 | 2
  Ptosis present, FE | 1 | 3 | 1 | 1 | 9 | 2 | 3
  2-step worsening of Meibomian gland dysfunction,SE | 0 | 0 | 2 | 0 | 2 | 0 | 0
  2-step worsening of Meibomian gland dysfunction,FE | 0 | 0 | 4 | 0 | 2 | 0 | 0
  2-step worsening of Conjunctival injection, SE | 2 | 0 | 1 | 0 | 1 | 5 | 0
  2-step worsening of Conjunctival injection, FE | 1 | 1 | 1 | 1 | 1 | 3 | 1
  2-step worsening of Chemosis, SE | 0 | 0 | 0 | 0 | 1 | 1 | 0
  2-step worsening of Chemosis, FE | 0 | 0 | 0 | 0 | 1 | 1 | 0
  2-step worsening of punctate keratopathy, SE | 0 | 0 | 1 | 0 | 2 | 4 | 0
  2-step worsening of punctate keratopathy, FE | 0 | 1 | 2 | 0 | 1 | 0 | 2
  2-step worsening of epithelial edema, SE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  2-step worsening of epithelial edema, FE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal postbaseline finding of active opacity,SE | 1 | 0 | 3 | 0 | 1 | 0 | 0
  Abnormal postbaseline finding of active opacity,FE | 2 | 0 | 3 | 0 | 2 | 0 | 0
  Abnormal post-baseline finding of active edema, SE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal post-baseline finding of active edema, FE | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1+ of Anterior chamber cell, SE | 0 | 1 | 0 | 1 | 1 | 0 | 1
  Grade 1+ of Anterior chamber cell, FE | 1 | 1 | 0 | 1 | 0 | 0 | 1
  Anterior chamber hypopyon present, SE | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Anterior chamber hypopyon present, FE | 0 | 0 | 2 | 2 | 0 | 0 | 0
  Grade 2+ of Anterior chamber flare, SE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2+ of Anterior chamber flare, FE | 0 | 0 | 0 | 1 | 0 | 0 | 0
  2+ increases in Any Lens Opacity, SE | 4 | 1 | 5 | 6 | 5 | 7 | 6
  2+ increases in Any Lens Opacity, FE | 3 | 1 | 4 | 4 | 4 | 4 | 6
  VA =>15 loss from Baseline or Previous Visit, SE | 15 | 8 | 7 | 9 | 9 | 16 | 5
  VA =>15 loss from Baseline or Previous Visit, FE | 10 | 5 | 6 | 10 | 5 | 5 | 6

13. Secondary Outcome: Summary of Intraocular Pressure Exam Findings
Description: Intraocular pressure (IOP) measurement was done with Goldmann tonometer. Intraocular pressure was measured prior to dilating the pupil and, to account for diurnal variation, at approximately the same time of day for every visit.
Time Frame: Up to week 52
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Participants
  Any post-baseline IOP >=30 study eye | 0 | 0 | 1 | 1 | 0 | 1 | 1
  IOP Lowering Medication for study eye | 1 | 4 | 5 | 6 | 4 | 3 | 6
  IOP Lowering procedure for study eye | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Any post-baseline IOP >=30 fellow eye | 0 | 0 | 0 | 1 | 0 | 0 | 2
  IOP Lowering Medication for fellow eye | 2 | 3 | 3 | 5 | 1 | 2 | 4
  IOP Lowering procedure for fellow eye | 1 | 1 | 1 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Vital Sign Values Outside of Clinical Concern Range
Description: Vital signs including systolic and diastolic blood pressure and heart rate were measured throughout the study. Number of participants with vital signs outside of clinical concern Range were summarized. 'High' denotes above normal range and 'Low' denotes below normal range for all the categories. The potential clinical importance ranges (low and high) of the vital sign parameters were for systolic blood pressure (<85 and >160 millimeter of mercury [mmHg]), diastolic blood pressure (<45 and >100 mmHg) and heart rate (<40 and >110 beats per minute). Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important vital parameter findings at any visit were reported.
Time Frame: Up to Week 52
Population: Safety Population. Only participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Participants
  Average diastolic blood pressure, Week 4, High: number analyzed (Participants) | 72 | 71 | 74 | 73 | 73 | 71 | 73
  Average diastolic blood pressure, Week 4, High | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Average diastolic blood pressure, Week 4, Low: number analyzed (Participants) | 72 | 71 | 74 | 73 | 73 | 71 | 73
  Average diastolic blood pressure, Week 4, Low | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Average diastolic blood pressure, Week 8, High: number analyzed (Participants) | 72 | 70 | 74 | 73 | 72 | 71 | 72
  Average diastolic blood pressure, Week 8, High | 1 | 0 | 0 | 0 | 1 | 1 | 0
  Average diastolic blood pressure, Week 12, High: number analyzed (Participants) | 72 | 68 | 74 | 73 | 72 | 71 | 69
  Average diastolic blood pressure, Week 12, High | 1 | 0 | 1 | 0 | 0 | 2 | 1
  Average diastolic blood pressure, Week 16, High: number analyzed (Participants) | 72 | 68 | 73 | 70 | 71 | 69 | 68
  Average diastolic blood pressure, Week 16, High | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Average diastolic blood pressure, Week 20, High: number analyzed (Participants) | 70 | 68 | 72 | 70 | 71 | 69 | 67
  Average diastolic blood pressure, Week 20, High | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Average diastolic blood pressure, Week 24, High: number analyzed (Participants) | 70 | 68 | 72 | 69 | 71 | 69 | 66
  Average diastolic blood pressure, Week 24, High | 0 | 0 | 1 | 0 | 1 | 1 | 0
  Average diastolic blood pressure, Week 24, Low: number analyzed (Participants) | 70 | 68 | 72 | 69 | 71 | 69 | 66
  Average diastolic blood pressure, Week 24, Low | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Average diastolic blood pressure, Week 28, Low: number analyzed (Participants) | 69 | 68 | 71 | 69 | 70 | 68 | 66
  Average diastolic blood pressure, Week 28, Low | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Average diastolic blood pressure, Week 32, High: number analyzed (Participants) | 68 | 68 | 70 | 69 | 68 | 67 | 62
  Average diastolic blood pressure, Week 32, High | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Average diastolic blood pressure, Week 36, Low: number analyzed (Participants) | 67 | 66 | 71 | 68 | 69 | 67 | 64
  Average diastolic blood pressure, Week 36, Low | 0 | 0 | 0 | 2 | 0 | 0 | 1
  Average diastolic blood pressure, Week 44, High: number analyzed (Participants) | 67 | 68 | 70 | 67 | 67 | 65 | 63
  Average diastolic blood pressure, Week 44, High | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Average diastolic blood pressure, Week 48, High: number analyzed (Participants) | 65 | 66 | 71 | 66 | 68 | 66 | 62
  Average diastolic blood pressure, Week 48, High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Average diastolic blood pressure, Week 52, High: number analyzed (Participants) | 65 | 66 | 71 | 67 | 67 | 64 | 62
  Average diastolic blood pressure, Week 52, High | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Average systolic blood pressure, Day 1, High | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Average systolic blood pressure, Week 4, High: number analyzed (Participants) | 72 | 71 | 74 | 73 | 73 | 71 | 73
  Average systolic blood pressure, Week 4, High | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Average systolic blood pressure, Week 8, High: number analyzed (Participants) | 72 | 70 | 74 | 73 | 72 | 71 | 72
  Average systolic blood pressure, Week 8, High | 0 | 1 | 0 | 1 | 0 | 1 | 1
  Average systolic blood pressure, Week 12, High: number analyzed (Participants) | 72 | 68 | 74 | 72 | 72 | 69 | 69
  Average systolic blood pressure, Week 12, High | 0 | 0 | 0 | 2 | 1 | 5 | 2
  Average systolic blood pressure, Week 16, High: number analyzed (Participants) | 72 | 68 | 73 | 70 | 71 | 69 | 68
  Average systolic blood pressure, Week 16, High | 0 | 1 | 0 | 1 | 2 | 1 | 2
  Average systolic blood pressure, Week 20, High: number analyzed (Participants) | 70 | 68 | 72 | 70 | 71 | 69 | 67
  Average systolic blood pressure, Week 20, High | 1 | 0 | 3 | 0 | 3 | 1 | 1
  Average systolic blood pressure, Week 24, High: number analyzed (Participants) | 70 | 68 | 72 | 69 | 71 | 69 | 66
  Average systolic blood pressure, Week 24, High | 0 | 0 | 3 | 1 | 3 | 1 | 2
  Average systolic blood pressure, Week 28, High: number analyzed (Participants) | 69 | 68 | 71 | 69 | 70 | 68 | 66
  Average systolic blood pressure, Week 28, High | 1 | 0 | 0 | 5 | 1 | 3 | 5
  Average systolic blood pressure, Week 32, High: number analyzed (Participants) | 68 | 68 | 70 | 69 | 68 | 67 | 62
  Average systolic blood pressure, Week 32, High | 0 | 0 | 2 | 0 | 1 | 2 | 0
  Average systolic blood pressure, Week 36, High: number analyzed (Participants) | 67 | 66 | 71 | 68 | 69 | 67 | 64
  Average systolic blood pressure, Week 36, High | 1 | 0 | 2 | 2 | 0 | 2 | 1
  Average systolic blood pressure, Week 40, High: number analyzed (Participants) | 68 | 68 | 70 | 68 | 67 | 67 | 63
  Average systolic blood pressure, Week 40, High | 1 | 0 | 2 | 1 | 0 | 1 | 1
  Average systolic blood pressure, Week 44, High: number analyzed (Participants) | 67 | 68 | 70 | 73 | 73 | 72 | 73
  Average systolic blood pressure, Week 44, High | 2 | 0 | 0 | 1 | 2 | 0 | 0
  Average systolic blood pressure, Week 44, Low: number analyzed (Participants) | 67 | 68 | 70 | 73 | 73 | 72 | 73
  Average systolic blood pressure, Week 44, Low | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Average systolic blood pressure, Week 48, High: number analyzed (Participants) | 65 | 66 | 71 | 73 | 73 | 72 | 73
  Average systolic blood pressure, Week 48, High | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Average systolic blood pressure, Week 52, High: number analyzed (Participants) | 65 | 66 | 71 | 73 | 73 | 72 | 73
  Average systolic blood pressure, Week 52, High | 2 | 2 | 2 | 1 | 2 | 2 | 2
  Heart Rate, Week 16, High: number analyzed (Participants) | 71 | 68 | 73 | 70 | 71 | 69 | 68
  Heart Rate, Week 16, High | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Heart Rate, Week 20, High: number analyzed (Participants) | 70 | 68 | 72 | 70 | 71 | 69 | 67
  Heart Rate, Week 20, High | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Heart Rate, Week 24, High: number analyzed (Participants) | 70 | 68 | 72 | 69 | 71 | 69 | 66
  Heart Rate, Week 24, High | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Heart Rate, Week 32, High: number analyzed (Participants) | 68 | 68 | 70 | 69 | 68 | 66 | 62
  Heart Rate, Week 32, High | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Heart Rate, Week 36, High: number analyzed (Participants) | 67 | 66 | 71 | 68 | 69 | 67 | 64
  Heart Rate, Week 36, High | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Heart Rate, Week 40, High: number analyzed (Participants) | 68 | 68 | 70 | 68 | 67 | 67 | 63
  Heart Rate, Week 40, High | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Heart Rate, Week 48, High: number analyzed (Participants) | 65 | 66 | 71 | 68 | 66 | 68 | 62
  Heart Rate, Week 48, High | 0 | 1 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Summary of Abnormal Electrocardiogram (ECG) Findings
Description: 12-Lead ECGs were performed in triplicate and were obtained on Weeks 4 to Week 28 and Week 52. The on-treatment ECGs were used to ascertain any risk of QTc interval prolongation at extremely low pazopanib exposures compared to what was routinely observed in participants with cancer. The on-treatment ECG data collected from participants assigned to one of the control arms also provided ECG background rate data for participants not exposed to pazopanib. Participants with Clinically significant abnormal ECGs are included here.
Time Frame: Week 4, Week 28, Week 44 and Week 52
Population: Safety population. Only participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Participants
  Week 4, Abnormal - Clinically significant: number analyzed (Participants) | 72 | 70 | 74 | 73 | 72 | 72 | 71
  Week 4, Abnormal - Clinically significant | 10 | 11 | 13 | 10 | 13 | 17 | 15
  Week 4, Abnormal - Not Clinically significant: number analyzed (Participants) | 72 | 70 | 74 | 73 | 72 | 72 | 71
  Week 4, Abnormal - Not Clinically significant | 24 | 25 | 25 | 25 | 24 | 31 | 27
  Week 28, Abnormal - Clinically significant: number analyzed (Participants) | 52 | 49 | 54 | 52 | 46 | 49 | 49
  Week 28, Abnormal - Clinically significant | 10 | 8 | 9 | 10 | 7 | 7 | 16
  Week 28, Abnormal - Not Clinically significant: number analyzed (Participants) | 52 | 49 | 54 | 52 | 46 | 49 | 49
  Week 28, Abnormal - Not Clinically significant | 21 | 22 | 17 | 22 | 18 | 25 | 18
  Week 44, Abnormal - Clinically significant: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Week 44, Abnormal - Clinically significant |  | 0 |  |  |  |  | 1
  Week 44, Abnormal - Not Clinically significant: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Week 44, Abnormal - Not Clinically significant |  | 1 |  |  |  |  | 0
  Week 52, Abnormal - Clinically significant: number analyzed (Participants) | 57 | 54 | 63 | 59 | 60 | 52 | 53
  Week 52, Abnormal - Clinically significant | 11 | 5 | 11 | 10 | 8 | 9 | 10
  Week 52, Abnormal - Not Clinically significant: number analyzed (Participants) | 57 | 54 | 63 | 59 | 60 | 52 | 53
  Week 52, Abnormal - Not Clinically significant | 23 | 29 | 25 | 21 | 24 | 22 | 20

16. Secondary Outcome: Summary of Hematology and Clinical Chemistry Parameters Data of Clinical Concern
Description: The Laboratory Parameters included Alanine Amino Transferase (ALT), Albumin, Alkaline Phosphatase, Aspartate Amino Transferase (AST), Calcium, Bicarbonate, Creatinine, Glucose, Hemoglobin, Lymphocytes, Platelet count, Potassium, Sodium, Thyroid Stimulating Hormone (TSH), Total Bilirubin, Total Neutrophils, Blood Urea Nitrogen (BUN) and White Blood Cell count (WBC). Number of participants with Laboratory outside of clinical concern Range were summarized here. Data of high and low from the clinical concern range has been provided here. Here 'High' denotes above normal range and 'Low' denotes below normal range for all the categories.
Time Frame: Up to Week 52
Population: Safety Population. Only participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Participants
  ALT, Week 4, High: number analyzed (Participants) | 71 | 70 | 72 | 70 | 71 | 70 | 73
  ALT, Week 4, High | 0 | 0 | 2 | 0 | 0 | 0 | 0
  ALT, Week 8, High: number analyzed (Participants) | 69 | 68 | 72 | 69 | 68 | 67 | 69
  ALT, Week 8, High | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALT, Week 12, High: number analyzed (Participants) | 70 | 67 | 71 | 70 | 70 | 67 | 65
  ALT, Week 12, High | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALT, Week 52, High: number analyzed (Participants) | 65 | 62 | 68 | 63 | 65 | 63 | 61
  ALT, Week 52, High | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Albumin, Week 4, Low: number analyzed (Participants) | 71 | 70 | 72 | 70 | 72 | 70 | 73
  Albumin, Week 4, Low | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, Week 12, High: number analyzed (Participants) | 70 | 67 | 71 | 70 | 70 | 67 | 65
  Alkaline Phosphatase, Week 12, High | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, Week 16, High: number analyzed (Participants) | 65 | 66 | 70 | 66 | 70 | 67 | 65
  Alkaline Phosphatase, Week 16, High | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, Week 20, High: number analyzed (Participants) | 68 | 66 | 72 | 70 | 70 | 69 | 64
  Alkaline Phosphatase, Week 20, High | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, Week 24, High: number analyzed (Participants) | 68 | 64 | 72 | 68 | 66 | 65 | 62
  Alkaline Phosphatase, Week 24, High | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Week 8, High: number analyzed (Participants) | 69 | 68 | 72 | 69 | 69 | 67 | 69
  AST, Week 8, High | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST, Week 12, High: number analyzed (Participants) | 70 | 67 | 70 | 69 | 70 | 66 | 65
  AST, Week 12, High | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST, Week 16, High: number analyzed (Participants) | 64 | 67 | 71 | 67 | 70 | 68 | 66
  AST, Week 16, High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  AST, Week 20, High: number analyzed (Participants) | 68 | 66 | 72 | 70 | 70 | 69 | 64
  AST, Week 20, High | 0 | 1 | 0 | 0 | 0 | 0 | 1
  AST, Week 48, High: number analyzed (Participants) | 65 | 64 | 66 | 63 | 64 | 63 | 62
  AST, Week 48, High | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Calcium, Day 1, High: number analyzed (Participants) | 72 | 70 | 70 | 69 | 63 | 70 | 71
  Calcium, Day 1, High | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Calcium, Week 4, High: number analyzed (Participants) | 71 | 70 | 72 | 70 | 72 | 70 | 73
  Calcium, Week 4, High | 1 | 0 | 0 | 1 | 1 | 0 | 0
  Calcium, Week 12, High: number analyzed (Participants) | 69 | 66 | 70 | 69 | 69 | 66 | 65
  Calcium, Week 12, High | 2 | 0 | 0 | 0 | 1 | 0 | 0
  Calcium, Week 28, High: number analyzed (Participants) | 67 | 65 | 67 | 67 | 68 | 65 | 63
  Calcium, Week 28, High | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Calcium, Week 52, Low: number analyzed (Participants) | 65 | 61 | 68 | 63 | 65 | 63 | 61
  Calcium, Week 52, Low | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Bicarbonate, Day 1, High: number analyzed (Participants) | 72 | 70 | 70 | 69 | 69 | 70 | 71
  Bicarbonate, Day 1, High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Bicarbonate, Week4, Low: number analyzed (Participants) | 71 | 70 | 72 | 70 | 71 | 70 | 73
  Bicarbonate, Week4, Low | 1 | 0 | 1 | 0 | 1 | 2 | 2
  Bicarbonate, Week 8, Low: number analyzed (Participants) | 1 | 1 | 1 | 2 | 0 | 1 | 2
  Bicarbonate, Week 8, Low | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Bicarbonate, Week 12, Low: number analyzed (Participants) | 69 | 66 | 70 | 69 | 69 | 66 | 65
  Bicarbonate, Week 12, Low | 0 | 1 | 1 | 1 | 2 | 1 | 1
  Bicarbonate, Week 28, Low: number analyzed (Participants) | 67 | 65 | 67 | 67 | 68 | 65 | 63
  Bicarbonate, Week 28, Low | 3 | 1 | 0 | 0 | 0 | 4 | 1
  Bicarbonate, Week 32, Low: number analyzed (Participants) | 1 | 1 | 2 | 0 | 0 | 2 | 1
  Bicarbonate, Week 32, Low | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Bicarbonate, Week 40, Low: number analyzed (Participants) | 65 | 63 | 68 | 65 | 68 | 65 | 62
  Bicarbonate, Week 40, Low | 0 | 1 | 1 | 1 | 0 | 1 | 1
  Bicarbonate, Week 52, Low: number analyzed (Participants) | 65 | 61 | 68 | 63 | 65 | 63 | 61
  Bicarbonate, Week 52, Low | 1 | 3 | 1 | 2 | 1 | 2 | 2
  Creatinine, Day 1, High: number analyzed (Participants) | 72 | 71 | 70 | 70 | 69 | 70 | 72
  Creatinine, Day 1, High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine, Week 4, High: number analyzed (Participants) | 71 | 70 | 72 | 70 | 72 | 70 | 73
  Creatinine, Week 4, High | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine, Week 12, High: number analyzed (Participants) | 69 | 66 | 71 | 70 | 70 | 67 | 65
  Creatinine, Week 12, High | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Creatinine, Week 28, High: number analyzed (Participants) | 67 | 66 | 69 | 67 | 68 | 65 | 63
  Creatinine, Week 28, High | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Creatinine, Week 52, High: number analyzed (Participants) | 65 | 62 | 68 | 62 | 66 | 63 | 61
  Creatinine, Week 52, High | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Glucose, Day 1, High: number analyzed (Participants) | 72 | 71 | 70 | 70 | 69 | 70 | 72
  Glucose, Day 1, High | 6 | 5 | 3 | 3 | 1 | 3 | 7
  Glucose, Day 1, Low: number analyzed (Participants) | 72 | 71 | 70 | 70 | 69 | 70 | 72
  Glucose, Day 1, Low | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Glucose, Week 4, High: number analyzed (Participants) | 71 | 70 | 72 | 70 | 72 | 70 | 73
  Glucose, Week 4, High | 2 | 3 | 3 | 4 | 2 | 2 | 3
  Glucose, Week 4, Low: number analyzed (Participants) | 71 | 70 | 72 | 70 | 72 | 70 | 73
  Glucose, Week 4, Low | 0 | 1 | 2 | 0 | 0 | 1 | 2
  Glucose, Week 8, High: number analyzed (Participants) | 1 | 1 | 1 | 2 | 0 | 1 | 2
  Glucose, Week 8, High | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Glucose, Week 12, High: number analyzed (Participants) | 69 | 66 | 71 | 70 | 70 | 67 | 65
  Glucose, Week 12, High | 3 | 5 | 3 | 2 | 4 | 2 | 8
  Glucose, Week 12, Low: number analyzed (Participants) | 69 | 66 | 71 | 70 | 70 | 67 | 65
  Glucose, Week 12, Low | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Glucose, Week 28, High: number analyzed (Participants) | 67 | 66 | 69 | 67 | 68 | 65 | 63
  Glucose, Week 28, High | 3 | 4 | 3 | 4 | 1 | 0 | 6
  Glucose, Week 28, Low: number analyzed (Participants) | 67 | 66 | 69 | 67 | 68 | 65 | 63
  Glucose, Week 28, Low | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Glucose, Week 32, High: number analyzed (Participants) | 1 | 1 | 2 | 0 | 1 | 2 | 1
  Glucose, Week 32, High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Glucose, Week 36, High: number analyzed (Participants) | 0 | 1 | 0 | 0 | 2 | 0 | 0
  Glucose, Week 36, High |  | 0 |  |  | 1 |  |
  Glucose, Week 40, High: number analyzed (Participants) | 65 | 63 | 68 | 65 | 68 | 65 | 62
  Glucose, Week 40, High | 6 | 7 | 4 | 5 | 1 | 3 | 9
  Glucose, Week 40, Low: number analyzed (Participants) | 65 | 63 | 68 | 65 | 68 | 65 | 62
  Glucose, Week 40, Low | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Glucose, Week 52, High: number analyzed (Participants) | 65 | 62 | 68 | 63 | 66 | 63 | 61
  Glucose, Week 52, High | 6 | 3 | 7 | 5 | 4 | 3 | 5
  Haemoglobin, Week 8, High: number analyzed (Participants) | 1 | 4 | 1 | 2 | 0 | 2 | 2
  Haemoglobin, Week 8, High | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes, Day 1, Low: number analyzed (Participants) | 69 | 70 | 72 | 71 | 70 | 70 | 72
  Lymphocytes, Day 1, Low | 1 | 3 | 3 | 3 | 3 | 0 | 1
  Lymphocytes, Week 4, Low: number analyzed (Participants) | 70 | 65 | 71 | 71 | 72 | 69 | 69
  Lymphocytes, Week 4, Low | 0 | 1 | 2 | 3 | 1 | 1 | 1
  Lymphocytes, Week 12, Low: number analyzed (Participants) | 70 | 64 | 71 | 69 | 71 | 68 | 66
  Lymphocytes, Week 12, Low | 2 | 0 | 2 | 2 | 2 | 2 | 1
  Lymphocytes, Week 28, Low: number analyzed (Participants) | 66 | 66 | 69 | 66 | 67 | 68 | 65
  Lymphocytes, Week 28, Low | 1 | 0 | 2 | 2 | 2 | 0 | 2
  Lymphocytes, Week 40, Low: number analyzed (Participants) | 64 | 64 | 66 | 67 | 68 | 63 | 62
  Lymphocytes, Week 40, Low | 2 | 1 | 3 | 4 | 0 | 1 | 0
  Lymphocytes, Week 52, Low: number analyzed (Participants) | 65 | 66 | 66 | 64 | 66 | 63 | 60
  Lymphocytes, Week 52, Low | 1 | 1 | 1 | 2 | 2 | 3 | 1
  Platelet count, Day 1, High: number analyzed (Participants) | 68 | 69 | 72 | 71 | 70 | 71 | 70
  Platelet count, Day 1, High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Platelet count, Day 1, Low: number analyzed (Participants) | 68 | 69 | 72 | 71 | 70 | 71 | 70
  Platelet count, Day 1, Low | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Platelet count, Week 4, High: number analyzed (Participants) | 69 | 64 | 69 | 70 | 72 | 67 | 71
  Platelet count, Week 4, High | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Platelet count, Week 4, Low: number analyzed (Participants) | 69 | 64 | 69 | 70 | 72 | 67 | 71
  Platelet count, Week 4, Low | 1 | 0 | 2 | 0 | 0 | 0 | 0
  Platelet count, Week 12, High: number analyzed (Participants) | 70 | 61 | 71 | 69 | 71 | 68 | 66
  Platelet count, Week 12, High | 1 | 0 | 0 | 1 | 0 | 2 | 0
  Platelet count, Week 12, Low: number analyzed (Participants) | 70 | 61 | 71 | 69 | 71 | 68 | 66
  Platelet count, Week 12, Low | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Platelet count, Week 28, High: number analyzed (Participants) | 64 | 66 | 68 | 66 | 67 | 68 | 65
  Platelet count, Week 28, High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Platelet count, Week 28, Low: number analyzed (Participants) | 64 | 66 | 68 | 66 | 67 | 68 | 65
  Platelet count, Week 28, Low | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Platelet count, Week 40, High: number analyzed (Participants) | 63 | 64 | 67 | 67 | 68 | 64 | 62
  Platelet count, Week 40, High | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Platelet count, Week 44, High: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 1 | 1
  Platelet count, Week 44, High | 0 | 0 |  |  |  | 1 | 0
  Platelet count, Week 52, High: number analyzed (Participants) | 65 | 66 | 67 | 66 | 66 | 62 | 60
  Platelet count, Week 52, High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Potassium, Day 1, High: number analyzed (Participants) | 72 | 70 | 70 | 69 | 69 | 70 | 71
  Potassium, Day 1, High | 1 | 3 | 1 | 0 | 0 | 0 | 0
  Potassium, Day 1, Low: number analyzed (Participants) | 72 | 70 | 70 | 69 | 69 | 70 | 71
  Potassium, Day 1, Low | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Potassium, Week 4, High: number analyzed (Participants) | 71 | 70 | 72 | 70 | 71 | 70 | 73
  Potassium, Week 4, High | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Potassium, Week 4, Low: number analyzed (Participants) | 71 | 70 | 72 | 70 | 71 | 70 | 73
  Potassium, Week 4, Low | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Potassium, Week 12, High: number analyzed (Participants) | 69 | 66 | 70 | 69 | 69 | 66 | 64
  Potassium, Week 12, High | 3 | 0 | 1 | 0 | 0 | 0 | 1
  Potassium, Week 12, Low: number analyzed (Participants) | 69 | 66 | 70 | 69 | 69 | 66 | 64
  Potassium, Week 12, Low | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Potassium, Week 28, High: number analyzed (Participants) | 67 | 65 | 67 | 67 | 68 | 65 | 63
  Potassium, Week 28, High | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Potassium, Week 40, High: number analyzed (Participants) | 65 | 63 | 68 | 65 | 68 | 65 | 62
  Potassium, Week 40, High | 0 | 1 | 0 | 2 | 0 | 1 | 0
  Potassium, Week 52, High: number analyzed (Participants) | 65 | 61 | 68 | 62 | 65 | 63 | 61
  Potassium, Week 52, High | 1 | 0 | 1 | 0 | 2 | 1 | 0
  Sodium, Week 12, High: number analyzed (Participants) | 69 | 66 | 71 | 70 | 70 | 67 | 65
  Sodium, Week 12, High | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, Week 40, Low: number analyzed (Participants) | 65 | 63 | 67 | 65 | 68 | 65 | 62
  Sodium, Week 40, Low | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Sodium, Week 52, Low: number analyzed (Participants) | 65 | 62 | 68 | 62 | 66 | 63 | 61
  Sodium, Week 52, Low | 0 | 0 | 0 | 0 | 0 | 0 | 2
  TSH, Day 1, High: number analyzed (Participants) | 59 | 62 | 63 | 63 | 59 | 64 | 61
  TSH, Day 1, High | 2 | 2 | 3 | 3 | 2 | 1 | 1
  TSH, Week 12, High: number analyzed (Participants) | 59 | 62 | 63 | 63 | 59 | 64 | 61
  TSH, Week 12, High | 1 | 1 | 2 | 1 | 1 | 3 | 0
  TSH, Week 24, High: number analyzed (Participants) | 64 | 64 | 66 | 62 | 59 | 59 | 58
  TSH, Week 24, High | 0 | 2 | 2 | 4 | 2 | 2 | 1
  TSH, Week 36, High: number analyzed (Participants) | 65 | 64 | 63 | 60 | 60 | 60 | 61
  TSH, Week 36, High | 1 | 2 | 3 | 5 | 3 | 2 | 2
  TSH, Week 52, High: number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 55 | 56
  TSH, Week 52, High | 3 | 2 | 1 | 4 | 2 | 3 | 4
  Total Bilirubin, Week 24, High: number analyzed (Participants) | 68 | 64 | 72 | 68 | 66 | 65 | 62
  Total Bilirubin, Week 24, High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Total Bilirubin, Week 32, High: number analyzed (Participants) | 67 | 64 | 66 | 64 | 66 | 65 | 61
  Total Bilirubin, Week 32, High | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, Week 44, High: number analyzed (Participants) | 62 | 63 | 69 | 65 | 65 | 61 | 60
  Total Bilirubin, Week 44, High | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Total Neutrophils, Day 1, Low: number analyzed (Participants) | 69 | 70 | 72 | 71 | 70 | 70 | 72
  Total Neutrophils, Day 1, Low | 0 | 1 | 2 | 0 | 1 | 0 | 2
  Total Neutrophils, Week 4, Low: number analyzed (Participants) | 70 | 65 | 71 | 71 | 72 | 69 | 69
  Total Neutrophils, Week 4, Low | 0 | 1 | 1 | 0 | 0 | 1 | 1
  Total Neutrophils, Week 12, Low: number analyzed (Participants) | 70 | 64 | 71 | 69 | 71 | 68 | 66
  Total Neutrophils, Week 12, Low | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Total Neutrophils, Week 32, Low: number analyzed (Participants) | 2 | 1 | 0 | 0 | 2 | 2 | 1
  Total Neutrophils, Week 32, Low | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Total Neutrophils, Week 40, Low: number analyzed (Participants) | 64 | 64 | 66 | 67 | 68 | 63 | 62
  Total Neutrophils, Week 40, Low | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Total Neutrophils, Week 52, Low: number analyzed (Participants) | 65 | 66 | 66 | 64 | 66 | 63 | 60
  Total Neutrophils, Week 52, Low | 0 | 0 | 0 | 0 | 1 | 0 | 0
  BUN, Day 1, High: number analyzed (Participants) | 72 | 71 | 70 | 70 | 69 | 70 | 72
  BUN, Day 1, High | 1 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, Week 4, High: number analyzed (Participants) | 71 | 70 | 72 | 70 | 72 | 70 | 73
  BUN, Week 4, High | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, Week 12, High: number analyzed (Participants) | 69 | 66 | 71 | 70 | 70 | 67 | 65
  BUN, Week 12, High | 0 | 0 | 0 | 1 | 0 | 2 | 1
  BUN, Week 16, High: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0 | 1
  BUN, Week 16, High | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BUN, Week 28, High: number analyzed (Participants) | 67 | 66 | 69 | 67 | 68 | 65 | 63
  BUN, Week 28, High | 0 | 0 | 0 | 0 | 0 | 0 | 1
  BUN, Week 40, High: number analyzed (Participants) | 65 | 63 | 68 | 65 | 68 | 65 | 62
  BUN, Week 40, High | 0 | 0 | 0 | 3 | 0 | 0 | 1
  WBC, DAy 1, Low: number analyzed (Participants) | 69 | 70 | 72 | 71 | 70 | 70 | 72
  WBC, DAy 1, Low | 0 | 1 | 1 | 0 | 0 | 0 | 0
  WBC, Week 28, Low: number analyzed (Participants) | 66 | 66 | 69 | 67 | 67 | 68 | 65
  WBC, Week 28, Low | 0 | 0 | 0 | 0 | 0 | 0 | 1
  WBC, Week 52, High: number analyzed (Participants) | 65 | 66 | 66 | 65 | 66 | 63 | 60
  WBC, Week 52, High | 1 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Laboratory Data of Clinical Concern for Urine Protein
Description: Urine Samples were collected from Day 1 to Week 28 and Week 52 for analyses. In this dipstick test, the level of protein in urine samples was recorded as negative (Neg), trace (tr), 1+, 2+, and 3+ (the plus sign increases with a higher level of proteins in the urine: 1+=slightly positive, 2+=positive, 3+=high positive). Neg indicated no proteinuria and 3+(high positive) indicated worst proteinuria.
Time Frame: Day 1 to Week 28 and Week 52
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
Number analyzed (Participants) | 73 | 72 | 74 | 73 | 73 | 72 | 73
Participants
  Week 4: number analyzed (Participants) | 71 | 68 | 72 | 67 | 72 | 69 | 72
  Week 4 | 7 | 3 | 5 | 6 | 2 | 1 | 2
  Week 8: number analyzed (Participants) | 1 | 1 | 2 | 2 | 0 | 3 | 3
  Week 8 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Week 16: number analyzed (Participants) | 1 | 0 | 2 | 0 | 0 | 0 | 0
  Week 16 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 61 | 68 | 70 | 68 | 69 | 66 | 62
  Week 28 | 7 | 5 | 4 | 8 | 4 | 2 | 6
  Week 32: number analyzed (Participants) | 3 | 2 | 0 | 0 | 2 | 2 | 1
  Week 32 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Week 52: number analyzed (Participants) | 60 | 64 | 69 | 65 | 66 | 64 | 59
  Week 52 | 2 | 3 | 8 | 10 | 5 | 3 | 3

18. Secondary Outcome: Plasma Concentrations of Pazopanib
Description: All participants in the eye drop containing arms had a single blood sample drawn for assessment of pazopanib plasma concentration at the Week 4, Week 24 and Week 24. The sample was drawn without restriction for the time interval between blood draw and the last dose of IP eye drops.
Time Frame: Week 4, Week 24 and Week 52
Population: Safety Population. Only participants with data available at the indicated time points were analyzed.
Measure: Mean (95% Confidence Interval); unit: nanogram/milliliter
Arm/Group | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID
Number analyzed (Participants) | 72 | 74 | 73 | 73 | 72
nanogram/milliliter
  Week 4: number analyzed (Participants) | 67 | 72 | 71 | 70 | 70
  Week 4 | 80.20 [64.66 to 95.74] | 103.38 [89.68 to 117.08] | 93.82 [72.51 to 115.13] | 114.33 [96.77 to 131.90] | 175.89 [148.80 to 202.98]
  Week 24: number analyzed (Participants) | 68 | 72 | 69 | 66 | 65
  Week 24 | 81.94 [67.45 to 96.44] | 101.96 [86.10 to 117.82] | 104.88 [73.09 to 136.68] | 114.58 [96.71 to 132.45] | 183.32 [146.70 to 219.94]
  Week 52: number analyzed (Participants) | 1 | 1 | 3 | 2 | 1
  Week 52 | NA [NA to NA] — NA indicates, data not quantifiable because the concentration was below limit of quantification. | 44.04 [NA to NA] — Only one participant was available at the time of analysis, confidence interval could not be calculated. | 60.98 [-79.29 to 201.25] | 28.77 [-227.64 to 285.18] | 40.33 [NA to NA] — Only one participant was available at the time of analysis, confidence interval could not be calculated.

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected during the treatment period (up to 52 weeks)
Description: All AEs and SAEs were reported on Safety Population.
Arm/Group | Placebo Control Arm QID | Pazopanib Eye Drops 5 mg/mL TID | Pazopanib Eye Drops 5 mg/mL QID | Pazopanib Eye Drops 10 mg/mL BID | Pazopanib Eye Drops 10 mg/mL TID | Pazopanib Eye Drops 10 mg/mL QID | Ranibizumab Injections Active Open-label Control Arm
All-Cause Mortality (participants affected / at risk) | 2/73 | 1/72 | 1/74 | 0/73 | 3/73 | 0/72 | 1/73
Serious Adverse Events (participants affected / at risk) | 11/73 | 10/72 | 12/74 | 11/73 | 10/73 | 11/72 | 6/73
Other Adverse Events (participants affected / at risk) | 52/73 | 34/72 | 47/74 | 44/73 | 46/73 | 41/72 | 42/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Control Arm QID (N=73) | Pazopanib Eye Drops 5 mg/mL TID (N=72) | Pazopanib Eye Drops 5 mg/mL QID (N=74) | Pazopanib Eye Drops 10 mg/mL BID (N=73) | Pazopanib Eye Drops 10 mg/mL TID (N=73) | Pazopanib Eye Drops 10 mg/mL QID (N=72) | Ranibizumab Injections Active Open-label Control Arm (N=73)
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain Stem Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device failure (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Control Arm QID (N=73) | Pazopanib Eye Drops 5 mg/mL TID (N=72) | Pazopanib Eye Drops 5 mg/mL QID (N=74) | Pazopanib Eye Drops 10 mg/mL BID (N=73) | Pazopanib Eye Drops 10 mg/mL TID (N=73) | Pazopanib Eye Drops 10 mg/mL QID (N=72) | Ranibizumab Injections Active Open-label Control Arm (N=73)
Nasopharyngitis (Infections and infestations) | 11 | 5 | 6 | 17 | 5 | 13 | 5
Hypertension (Vascular disorders) | 3 | 4 | 5 | 4 | 6 | 6 | 7
Urinary tract infection (Infections and infestations) | 9 | 3 | 1 | 6 | 6 | 4 | 3
Conjunctival haemorrhage (Eye disorders) | 5 | 2 | 1 | 7 | 6 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 6 | 4 | 2 | 3 | 3
Headache (Nervous system disorders) | 3 | 2 | 1 | 5 | 5 | 7 | 6
Retinal haemorrhage (Eye disorders) | 5 | 3 | 3 | 2 | 4 | 3 | 4
Visual acuity reduced (Eye disorders) | 3 | 3 | 2 | 1 | 6 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5 | 2 | 4 | 2 | 1
Eye pain (Eye disorders) | 7 | 1 | 1 | 1 | 4 | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 6 | 2 | 4 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 2 | 5 | 2 | 3 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 4 | 3 | 1 | 4 | 5
Vitreous floaters (Eye disorders) | 3 | 2 | 2 | 3 | 2 | 3 | 4
Bronchitis (Infections and infestations) | 3 | 1 | 2 | 2 | 4 | 2 | 4
Vision blurred (Eye disorders) | 4 | 1 | 2 | 2 | 4 | 2 | 2
Influenza (Infections and infestations) | 0 | 5 | 2 | 3 | 3 | 0 | 3
Pain (General disorders) | 1 | 4 | 2 | 3 | 2 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4 | 2 | 2 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 3 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2 | 0 | 3 | 4
Blepharitis (Eye disorders) | 2 | 0 | 3 | 1 | 3 | 0 | 4
Fall (Injury, poisoning and procedural complications) | 2 | 4 | 2 | 2 | 2 | 1 | 0
Punctate keratitis (Eye disorders) | 4 | 1 | 0 | 1 | 3 | 3 | 1
Seasonal allergy (Immune system disorders) | 3 | 1 | 4 | 2 | 0 | 1 | 2
Lacrimation increased (Eye disorders) | 0 | 1 | 1 | 2 | 1 | 5 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 5 | 3
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 4 | 2 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 2 | 0 | 1 | 6 | 0
Dry eye (Eye disorders) | 1 | 1 | 1 | 0 | 1 | 4 | 1
Injection site haemorrhage (General disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 4
Pneumonia (Infections and infestations) | 2 | 0 | 4 | 3 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 4 | 1 | 0 | 0 | 2
Cataract cortical (Eye disorders) | 1 | 0 | 4 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.